CLINICAL TRIAL: NCT04760873
Title: Gastric Antral Vascular Ectasia Treatment With Balloon Cryotherapy: A Multicenter Prospective Trial
Brief Title: Cryotherapy for GAVE
Acronym: GAVE Cryo
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal Investigator has not current plans or ability to mov the Study forward.
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Long Island Jewish Medical Center (Other); Geisinger Clinic (Other); Columbia University (Other); University Hospitals Cleveland Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-21904
Record Dates: First submitted 2021-02-15; First posted 2021-02-18 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: GAVE - Gastric Antral Vascular Ectasia; Bleeding; Bleeding Gastric
Keywords: GAVE; cryotherapy; bleeding; stomach; gastric; EGD; endoscopy
MeSH Terms: conditions — Gastric Antral Vascular Ectasia; Hemorrhage | interventions — Cryotherapy

STUDY DESIGN:
Intervention Model Description: Subjects with GAVE will undergo therapy with a cryotherapy device
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Cryotherapy for GAVE (Experimental): Subjects will undergo cryotherapy for GAVE
  Interventions: Device: cryotherapy

INTERVENTIONS:
Device: cryotherapy — cryotherapy is a freeze spray that will be applied to GAVE for bleeding

SUMMARY:
Gastric antral vascular ectasia (GAVE) is a condition that can lead to blood loss in the gastrointestinal tract and low blood counts or anemia. 1,2 GAVE is commonly associated with liver disease, kidney disease and autoimmune immune problems, but can also be seen in patients without those problems. 2-4 It is common for GAVE to cause hospitalization of patients and significant blood transfusion requirements. Given these problems, effective treatment of GAVE is needed to reduce these potential problems.

These treatments are performed by a gastroenterologist through a flexible endoscope most often with argon plasma coagulation (APC).5-7 APC is only partially successful at eradicating GAVE and often entails repeated endoscopic procedures. Therapy with APC can also cause ulceration at times resulting in acute bleeding. Cryoablation is an attractive alternative to APC as it should not cause increased blood loss and case reports suggest that ablation may be achieved with limited number of endoscopic sessions. Prior problems with endoscopic cryotherapy include the high flow of gas and risk of perforation.8,9 A recent retrospective investigation by this group has evaluated the first generation cryotherapy balloon, demonstrating clinical safety and efficacy for GAVE.10 A new balloon cryotherapy spray device was recently developed and does not require venting. In this study we plan to prospectively evaluate the use of balloon cryotherapy to treat GAVE. We predict that the therapeutic response of balloon cryotherapy will be greater than 80% effective at achieving clinical success or the loss of overt bleeding and need for packed red blood cell (PRBC) transfusion at 6 months after treatment.

DETAILED DESCRIPTION:
Gastric antral vascular ectasia (GAVE), classically termed "watermelon stomach," is a condition of chronic acute blood loss in the gastrointestinal (GI) tract and can lead to common utilization of packed red blood cell (PRBC) transfusion. This condition occurs in 0.3% of endoscopic studies and 4% of studies performed for chronic or acute blood loss anemia.1,2 GAVE is commonly associated with autoimmune disease in 60% of cases and chronic liver disease in 30% of cases.2-4 Given the association with chronic liver disease, GAVE can be mistaken for other GI pathologies such as portal hypertensive gastropathy (PHG).11,12 Therefore, identification of GAVE is important in the management of this condition.

Historically there have been 1 series highlighting the use of a monopolar probe and heater probe to treat GAVE. As these therapies have a low depth of thermal penetration, these therapies are not commonly utilized for GAVE.13,14 The most commonly implemented endoscopic therapy is argon plasma coagulation (APC). Among the largest studies of APC, the efficacy for treatment of GAVE is variable5,6 Additional outcomes include a reduction in the number of PRBC transfused in patients with GAVE that were treated with APC.7 In addition to APC, radiofrequency ablation (RFA) has also been evaluated in the setting of GAVE, leading to a decrease in the transfusions needed during follow-up.15 Similarly, cryotherapy using a spray catheter has been evaluated for GAVE.8,9 In these studies, the patients did demonstrate endoscopic improvement, lower transfusion requirements, and normalization of their hemoglobin. Despite, these results, the spray cryotherapy device requires the use of a venting tube to prevent complications and carries with it technical limitations that can make ablation difficult. Our study group, which includes University Hospitals, Case Western Reserve, Long Island Jewish Medical Center, Geisinger Medical Center, Columbia University Medical Center and The Cleveland Clinic Foundation of America This group has recently evaluated the first generation balloon cryotherapy device for GAVE, demonstrating efficacy and safety.10 Therefore, in this study we set out to prospectively evaluate the efficacy of a new balloon cryotherapy device for the treatment of GAVE. We predict that balloon cryotherapy will lead to greater than 80% clinical success (need for PRBC transfusion and absent overt bleeding).

ELIGIBILITY:
Inclusion Criteria:

1. Have GAVE
2. Have had treatment discussion with non-study team member (physician or GI advanced practice provider) of alternatives and have elected Cryotherapy
3. Patients with signs of GI bleeding defined as hemoglobin drop > 2 grams/dL, need for PRBC transfusion or overt bleeding (melena, hematemesis, hematochezia)
4. Patients undergoing EGD with Ablation for GAVE (treatment naïve, RFA, banding, APC failures)
5. Patients who underwent their last ablation at least 4 weeks prior
6. Platelet count > 40,000
7. International normalized ratio (INR) < 1.5
8. Age > 18 years and < 90 years

Exclusion Criteria:

1. Age < 18 years OR > 90 years
2. Inability to obtain consent
3. Anticoagulants or anti-platelet agents use (excluding aspirin) within the last 7-10 days
4. Platelet count < 40,000
5. INR > 1.5

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-10-14 (Actual); Primary Completion 2024-01-22 (Actual); Study Completion 2024-01-22 (Actual)

PRIMARY OUTCOMES:
Clinical success | 6 months
  defined by the absence of PRBC transfusions and clinical evidence of bleeding

SECONDARY OUTCOMES:
Technical success | 6 months
  defined as the ability to treat > 75% of the endoscopic area
Endoscopic success | 6 months
  defined as resolution of > 75% of the visible GAVE endoscopic surface
Mean/total number of PRBC transfused | 6 months
  transfusion of packed red blood cells
Change in hemoglobin | 6 months
  change in the lab test hemoglobin in grams/deciLiter
Technical failure | 6 months
  defined as the need for additional ablative modalities to achieve the primary study outcome

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Columbia University Medical Center-NYPH, New York, New York
  - Cleveland Clinic Foundation of America, Cleveland, Ohio
  - Geisinger Medical Center, Danville, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Electronic health records database will allow for availability of demographic data and office-based follow-up records. ProVation MD software information will provide details regarding endoscopic parameters and intervention performed.
  Electronic records gathered for study purposes will only be available to study investigators and will be stored on an encrypted hard drive on a computer. Data will initially be entered with PHI attached so that all information can be obtained. Once all data collection is complete identifiers will be removed and random number assigned to the patients.
  Paper copies of study consents will be filled out in the endoscopy center and stored in a locked cabinet in the endoscopy center workroom. The door to the workroom with the cabinet is locked after hours and the endoscopy center is locked after hours as well.
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Background] Dulai GS, Jensen DM, Kovacs TO, Gralnek IM, Jutabha R. Endoscopic treatment outcomes in watermelon stomach patients with and without portal hypertension. Endoscopy. 2004 Jan;36(1):68-72. doi: 10.1055/s-2004-814112. PMID 14722858
- [Background] Jabbari M, Cherry R, Lough JO, Daly DS, Kinnear DG, Goresky CA. Gastric antral vascular ectasia: the watermelon stomach. Gastroenterology. 1984 Nov;87(5):1165-70. PMID 6332757
- [Background] Lee FI, Costello F, Flanagan N, Vasudev KS. Diffuse antral vascular ectasia. Gastrointest Endosc. 1984 Apr;30(2):87-90. doi: 10.1016/s0016-5107(84)72326-1. No abstract available. PMID 6714608
- [Background] Tobin RW, Hackman RC, Kimmey MB, Durtschi MB, Hayashi A, Malik R, McDonald MF, McDonald GB. Bleeding from gastric antral vascular ectasia in marrow transplant patients. Gastrointest Endosc. 1996 Sep;44(3):223-9. doi: 10.1016/s0016-5107(96)70155-4. PMID 8885337
- [Background] Roman S, Saurin JC, Dumortier J, Perreira A, Bernard G, Ponchon T. Tolerance and efficacy of argon plasma coagulation for controlling bleeding in patients with typical and atypical manifestations of watermelon stomach. Endoscopy. 2003 Dec;35(12):1024-8. doi: 10.1055/s-2003-44594. PMID 14648415
- [Background] Yusoff I, Brennan F, Ormonde D, Laurence B. Argon plasma coagulation for treatment of watermelon stomach. Endoscopy. 2002 May;34(5):407-10. doi: 10.1055/s-2002-25287. PMID 11972274
- [Background] Wahab PJ, Mulder CJ, den Hartog G, Thies JE. Argon plasma coagulation in flexible gastrointestinal endoscopy: pilot experiences. Endoscopy. 1997 Mar;29(3):176-81. doi: 10.1055/s-2007-1004159. PMID 9201466
- [Background] Kantsevoy SV, Cruz-Correa MR, Vaughn CA, Jagannath SB, Pasricha PJ, Kalloo AN. Endoscopic cryotherapy for the treatment of bleeding mucosal vascular lesions of the GI tract: a pilot study. Gastrointest Endosc. 2003 Mar;57(3):403-6. doi: 10.1067/mge.2003.115. PMID 12612530
- [Background] Cho S, Zanati S, Yong E, Cirocco M, Kandel G, Kortan P, May G, Marcon N. Endoscopic cryotherapy for the management of gastric antral vascular ectasia. Gastrointest Endosc. 2008 Nov;68(5):895-902. doi: 10.1016/j.gie.2008.03.1109. Epub 2008 Jul 21. PMID 18640673
- [Background] Patel AA, Trindade AJ, Diehl DL, Khara HS, Lee TP, Lee C, Sethi A. Nitrous oxide cryotherapy ablation for refractory gastric antral vascular ectasia. United European Gastroenterol J. 2018 Oct;6(8):1155-1160. doi: 10.1177/2050640618783537. Epub 2018 Jun 12. PMID 30288277
- [Background] RIDER JA, KLOTZ AP, KIRSNER JB. Gastritis with veno-capillary ectasia as a source of massive gastric hemorrhage. Gastroenterology. 1953 May;24(1):118-23. No abstract available. PMID 13052170
- [Background] Selinger CP, Ang YS. Gastric antral vascular ectasia (GAVE): an update on clinical presentation, pathophysiology and treatment. Digestion. 2008;77(2):131-7. doi: 10.1159/000124339. Epub 2008 Apr 4. PMID 18391491
- [Background] Petrini JL Jr, Johnston JH. Heat probe treatment for antral vascular ectasia. Gastrointest Endosc. 1989 Jul-Aug;35(4):324-8. doi: 10.1016/s0016-5107(89)72802-9. PMID 2788591
- [Background] Gross SA, Al-Haddad M, Gill KR, Schore AN, Wallace MB. Endoscopic mucosal ablation for the treatment of gastric antral vascular ectasia with the HALO90 system: a pilot study. Gastrointest Endosc. 2008 Feb;67(2):324-7. doi: 10.1016/j.gie.2007.09.020. PMID 18226696
- [Background] Yao K. The endoscopic diagnosis of early gastric cancer. Ann Gastroenterol. 2013;26(1):11-22. PMID 24714327
- [Background] Rey JF, Lambert R; ESGE Quality Assurance Committee. ESGE recommendations for quality control in gastrointestinal endoscopy: guidelines for image documentation in upper and lower GI endoscopy. Endoscopy. 2001 Oct;33(10):901-3. doi: 10.1055/s-2001-42537. No abstract available. PMID 11605605
- [Background] Scholvinck DW, Kunzli HT, Kestens C, Siersema PD, Vleggaar FP, Canto MI, Cosby H, Abrams JA, Lightdale CJ, Tejeda-Ramirez E, DeMeester SR, Greene CL, Jobe BA, Peters J, Bergman JJ, Weusten BL. Treatment of Barrett's esophagus with a novel focal cryoablation device: a safety and feasibility study. Endoscopy. 2015 Dec;47(12):1106-12. doi: 10.1055/s-0034-1392417. Epub 2015 Jul 9. PMID 26158241
- [Background] Cotton PB, Eisen GM, Aabakken L, Baron TH, Hutter MM, Jacobson BC, Mergener K, Nemcek A Jr, Petersen BT, Petrini JL, Pike IM, Rabeneck L, Romagnuolo J, Vargo JJ. A lexicon for endoscopic adverse events: report of an ASGE workshop. Gastrointest Endosc. 2010 Mar;71(3):446-54. doi: 10.1016/j.gie.2009.10.027. No abstract available. PMID 20189503